CLINICAL TRIAL: NCT01736826
Title: Comparative Study of Plasma Free DNA and Nucleosome Concentrations: Pathological Versus Normal Pregnancies
Brief Title: Free DNA and Nucleosome Concentrations in Pathological Pregnancies
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2012/SB-01; 2014-A01120-47 (Other: ANSM)
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2019-01

CONDITIONS: Pregnancy; Venous Thrombosis; Pulmonary Embolism; Hypertension, Pregnancy-Induced; Eclampsia; HELLP Syndrome; Pre-Eclampsia; Fetal Death; Placental Insufficiency
Keywords: plasma nucleosome concentration; plasma free DNA concentration
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Hypertension, Pregnancy-Induced; Eclampsia; HELLP Syndrome; Pre-Eclampsia; Fetal Death; Placental Insufficiency | interventions — BaseLine dental cement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At each visit a total of 36 ml of blood will be drawn (5 x EDTA tube = 5 x 4.5ml; 2 x CTAD tube = 2 x 4.5 ml and 1 dry tube = 4.5 ml).
  Tubes will be rapidly conditioned and samples stored at -80°C. After analysis, remaining samples will be stored in the Nîmes University Hospital Biological Collections.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Group P: pregnancy w/complications: The patient is pregnant and has complications typical of placental vascular disease (preeclampsia, eclampsia, HELLP syndrome, retro-placental hematoma, in utero fetal death) or venous thromboembolism (deep vein thrombosis, pulmonary embolism).
  100 patients will be included.
  Interventions to be administered: Bloodwork, baseline
  Interventions: Biological: Bloodwork, baseline
- Group T1: Healthy volunteers: Healthy volunteers with no history of chronic or neoplastic disease.
  30 healthy volunteers will be included.
  Interventions to be administered: Bloodwork, baseline
  Interventions: Biological: Bloodwork, baseline
- Group T2: Pregnancy, no complications: Pregnant patients with no identifiable pregnancy complications, and no history of chronic or neoplastic disease.
  50 pregnant volunteers will be included.
  Interventions to be administered: Bloodwork, baseline
  Interventions: Biological: Bloodwork, baseline
- Group T1x: 15 Healthy volunteers: 15 Healthy volunteers selected from group T1 (the first 15). These patients will have 2 additional months of follow up.
  Interventions to be administered: Blood work, Months 1 & 2
  Interventions: Biological: Bloodwork, baseline; Biological: Blood work, Months 1 & 2
- Group T2x: 15 Pregnancy, no complications: 15 patients selected from group T2 (the first 15); these patients will have 7 months of follow up during pregnancy.
  Interventions to be administered: Bloodwork, Months -1 to -6
  Interventions: Biological: Bloodwork, baseline; Biological: Bloodwork, Months -1 to -6

INTERVENTIONS:
Biological: Bloodwork, baseline — 36 ml of blood are drawn at baseline (last month of pregnancy for groups P and T2, inclusion for group T1) in order to quantify the following: plasma free DNA concentration, plasma nucleosome concentration, hemoglobin, platelets, leukocytes, polynuclear neutrophils, mean corpuscular volume, monocytes, mean corpuscular hemoglobin, lymphocytes, polynuclear eosinophils, polynuclear basophils, D-Dimers, Fibrin monomers, Trophoblast microparticles, Angiogenic marker CD146.
Biological: Blood work, Months 1 & 2 — 36 ml of blood are drawn at 1 & 2 months after inclusion in order to quantify the following: plasma free DNA concentration, plasma nucleosome concentration, hemoglobin, platelets, leukocytes, polynuclear neutrophils, mean corpuscular volume, monocytes, mean corpuscular hemoglobin, lymphocytes, polynuclear eosinophils, polynuclear basophils, D-Dimers, Fibrin monomers, Trophoblast microparticles, Angiogenic marker CD146.
  Groups: Group T1x: 15 Healthy volunteers
Biological: Bloodwork, Months -1 to -6 — 36 ml of blood are drawn at the third, fourth, fifth, sixth, seventh and eight months of normal pregnancy (corresponding to months -1 to -6 before comparative baseline; this group is included in the study early during pregnancy)in order to quantify the following: plasma free DNA concentration, plasma nucleosome concentration, hemoglobin, platelets, leukocytes, polynuclear neutrophils, mean corpuscular volume, monocytes, mean corpuscular hemoglobin, lymphocytes, polynuclear eosinophils, polynuclear basophils, D-Dimers, Fibrin monomers, Trophoblast microparticles, Angiogenic marker CD146.
  Groups: Group T2x: 15 Pregnancy, no complications

SUMMARY:
The primary objective of this study is to demonstrate that plasma concentrations of nucleosomes and free DNA differ between three groups:

1. pregnant patients with complications typical of placental insufficiency or venous thrombosis (group P),
2. healthy women (Group T1) and
3. healthy pregnant women (Group T2).

DETAILED DESCRIPTION:
Our secondary objectives include the following:

1. To describe, in 15 healthy, non-pregnant women changes in plasma concentrations of nucleosomes and free DNA over 3 months.
2. To describe, in 15 pregnant women (without complications), changes in plasma concentrations of nucleosomes and free DNA over the last 7 months of pregnancy
3. To show that plasma concentrations of nucleosomes and free DNA, in patients with complicated pregnancies differ according to the nature of the complication
4. To show that a relationship exists between the concentrations of nucleosomes, free DNA, and total granulocyte microparticles (and trophoblast particles for pregnant women)
5. To evaluate the relationship between nucleosome concentrations, free DNA concentrations and circulating leukocyte populations
6. To evaluate the relationship between nucleosome concentrations, free DNA concentrations and hemostasis markers
7. To describe changes in hemostasis markers throughout pregnancy
8. To evaluate the relationship between nucleosome concentrations, free DNA concentrations and the angiogenic marker CD146
9. To add to the Nîmes University Hospital biological collections.

ELIGIBILITY:
Inclusion Criteria for all patients:

* The patient must have given her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan

Inclusion Criteria for patients in group P:

* The patient is pregnant and has complications typical of placental vascular disease (preeclampsia, eclampsia, HELLP syndrome, retro-placental hematoma, in utero fetal death) or venous thromboembolism (deep vein thrombosis, pulmonary embolism)

Inclusion Criteria for patients in group T1:

* The patient is available for 3 months of follow-up
* The patient is a non-pregnant healthy volunteer
* No identifiable chronic pathologies
* No history of neoplastic disease
* No history of chronic infectious disease
* No acute disease (such as benign infection), now or within the past two weeks

Inclusion Criteria for patients in group T2:

* The patient is available for 7 months of follow-up
* The patient is pregnant, with no identifiable pregnancy complications
* No identifiable chronic pathologies
* No history of neoplastic disease
* No history of chronic infectious disease
* No acute disease (such as benign infection), now or within the past two weeks

Exclusion Criteria for all patients:

* The patient is participating in another study (with the exception of the following studies: PAPILLO-PMA (2013-A00538-37), ElastoMAP (2013-A01148-37), ElastoDéclenche (2014-A00828-39), LXRs (2009-A00968-49), Bakri (2013-A00914-41), OASIS 2 (2013-A00022-43)).
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient cannot read French
* The patient is receiving hormonal ovarian stimulation in the context of medically assisted procreation
* Impossible to perform venipuncture under good conditions
* New complication or pathology during the study (except for pregnancy complications in group P)

Exclusion Criteria for group P:

* Twin or multiple pregnancy
* The patient is participating in another study (with the exception of those mentioned in the exclusion criteria for all patients and the DG Postpartum study (2013-A00277-38)

Exclusion Criteria for group T1:

* The patient is pregnant
* The patient is breast feeding
* The patient has given birth within the last 3 months
* Known history of chronic disease
* History of treated neoplastic disease
* Acute disease within the past two weeks (includes benign disease)

Exclusion Criteria for group T2:

* Pregnancy with complications
* Known history of chronic disease
* History of treated neoplastic disease
* Acute disease within the past two weeks (includes benign disease)
* Twin or multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes three groups:
  Group P: 100 pregnant women with complications typical of placental vascular disease or venous thromboembolism.
  Group T1: 30 non-pregnant, healthy volunteers
  * The first 15 patients from group T1 will form group T1x. The latter group has two months of additional follow up.
  Group T2: 50 pregnant, healthy volunteers
  * The first 15 patients from group T2 will form group T2x. The latter group has 7 months of follow-up during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2015-06; Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Total plasma concentration of free DNA (ng/ml) | Base line (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Total plasma concentration of nucleosomes (AU) | Base line (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth

SECONDARY OUTCOMES:
Hemoglobin (g/l) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Platelets (g/l) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Leukocytes (g/l) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Polynuclear neutrophils(g/l) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Mean corpuscular volume (fL) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Monocytes (g/l) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Mean corpuscular hemoglobin (pg/GR) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Lymphocytes (g/l) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Polynuclear eosinophils (g/l) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Polynuclear basophils (g/l) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
D-dimers (ng/ml) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Fibrin monomers (ng/ml) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Trophoblast microparticles (%) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Angiogenic marker CD146 (ng/ml) | baseline (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Hemoglobin (g/l) | 1 month
  For group T1x only
Platelets (g/l) | 1 month
  For group T1x only
Leukocytes (g/l) | 1 month
  For group T1x only
Polynuclear neutrophils(g/l) | 1 month
  For group T1x only
Mean corpuscular volume (fL) | 1 month
  For group T1x only
Monocytes (g/l) | 1 month
  For group T1x only
Mean corpuscular hemoglobin (pg/GR) | 1 month
  For group T1x only
Lymphocytes (g/l) | 1 month
  For group T1x only
Polynuclear eosinophils (g/l) | 1 month
  For group T1x only
Polynuclear basophils (g/l) | 1 month
  For group T1x only
D-dimers (ng/ml) | 1 month
  For group T1x only
Fibrin monomers (ng/ml) | 1 month
  For group T1x only
Trophoblast microparticles (%) | 1 month
  For group T1x only
Angiogenic marker CD146 (ng/ml) | 1 month
  For group T1x only
Total plasma concentration of free DNA (ng/ml) | 1 month
  For group T1x only
Total plasma concentration of nucleosomes (AU) | 1 month
  For group T1x only
Hemoglobin (g/l) | 2 months
  For group T1x only
Platelets (g/l) | 2 months
  For group T1x only
Leukocytes (g/l) | 2 months
  For group T1x only
Polynuclear neutrophils(g/l) | 2 months
  For group T1x only
Mean corpuscular volume (fL) | 2 months
  For group T1x only
Monocytes (g/l) | 2 months
  For group T1x only
Mean corpuscular hemoglobin (pg/GR) | 2 months
  For group T1x only
Lymphocytes (g/l) | 2 months
  For group T1x only
Polynuclear eosinophils (g/l) | 2 months
  For group T1x only
Polynuclear basophils (g/l) | 2 months
  For group T1x only
D-dimers (ng/ml) | 2 months
  For group T1x only
Fibrin monomers (ng/ml) | 2 months
  For group T1x only
Trophoblast microparticles (%) | 2 months
  For group T1x only
Angiogenic marker CD146 (ng/ml) | 2 months
  For group T1x only
Total plasma concentration of free DNA (ng/ml) | 2 months
  For group T1x only
Total plasma concentration of nucleosomes (AU) | 2 months
  For group T1x only
Hemoglobin (g/l) | -1 months
  For group T2x only
Hemoglobin (g/l) | -2 months
  For group T2x only
Hemoglobin (g/l) | -3 months
  For group T2x only
Hemoglobin (g/l) | -4 months
  For group T2x only
Hemoglobin (g/l) | -5 months
  For group T2x only
Hemoglobin (g/l) | -6 months
  For group T2x only
Platelets (g/l) | -1 months
  For group T2x only
Platelets (g/l) | -2 months
  For group T2x only
Platelets (g/l) | -3 months
  For group T2x only
Platelets (g/l) | -4 months
  For group T2x only
Platelets (g/l) | -5 months
  For group T2x only
Platelets (g/l) | -6 months
  For group T2x only
Leukocytes (g/l) | -1 months
  For group T2x only
Leukocytes (g/l) | -2 months
  For group T2x only
Leukocytes (g/l) | -3 months
  For group T2x only
Leukocytes (g/l) | -4 months
  For group T2x only
Leukocytes (g/l) | -5 months
  For group T2x only
Leukocytes (g/l) | -6 months
  For group T2x only
Polynuclear neutrophils(g/l) | -1 months
  For group T2x only
Polynuclear neutrophils(g/l) | -2 months
  For group T2x only
Polynuclear neutrophils(g/l) | -3 months
  For group T2x only
Polynuclear neutrophils(g/l) | -4 months
  For group T2x only
Polynuclear neutrophils(g/l) | -5 months
  For group T2x only
Polynuclear neutrophils(g/l) | -6 months
  For group T2x only
Mean corpuscular volume (fL) | -1 months
  For group T2x only
Mean corpuscular volume (fL) | -2 months
  For group T2x only
Mean corpuscular volume (fL) | -3 months
  For group T2x only
Mean corpuscular volume (fL) | -4 months
  For group T2x only
Mean corpuscular volume (fL) | -5 months
  For group T2x only
Mean corpuscular volume (fL) | -6 months
  For group T2x only
Monocytes (g/l) | -1 months
  For group T2x only.
Monocytes (g/l) | -2 months
  For group T2x only.
Monocytes (g/l) | -3 months
  For group T2x only.
Monocytes (g/l) | -4 months
  For group T2x only.
Monocytes (g/l) | -5 months
  For group T2x only.
Monocytes (g/l) | -6 months
  For group T2x only.
Mean corpuscular hemoglobin (pg/GR) | -1 months
  For group T2x only.
Mean corpuscular hemoglobin (pg/GR) | -2 months
  For group T2x only.
Mean corpuscular hemoglobin (pg/GR) | -3 months
  For group T2x only.
Mean corpuscular hemoglobin (pg/GR) | -4 months
  For group T2x only.
Mean corpuscular hemoglobin (pg/GR) | -5 months
  For group T2x only.
Mean corpuscular hemoglobin (pg/GR) | -6 months
  For group T2x only.
Lymphocytes (g/l) | -1 months
  For group T2x only.
Lymphocytes (g/l) | -2 months
  For group T2x only.
Lymphocytes (g/l) | -3 months
  For group T2x only.
Lymphocytes (g/l) | -4 months
  For group T2x only.
Lymphocytes (g/l) | -5 months
  For group T2x only.
Lymphocytes (g/l) | -6 months
  For group T2x only.
Polynuclear eosinophils (g/l) | -1 months
  For group T2x only.
Polynuclear eosinophils (g/l) | -2 months
  For group T2x only.
Polynuclear eosinophils (g/l) | -3 months
  For group T2x only.
Polynuclear eosinophils (g/l) | -4 months
  For group T2x only.
Polynuclear eosinophils (g/l) | -5 months
  For group T2x only.
Polynuclear eosinophils (g/l) | -6 months
  For group T2x only.
Polynuclear basophils (g/l) | -1 months
  For group T2x only.
Polynuclear basophils (g/l) | -2 months
  For group T2x only.
Polynuclear basophils (g/l) | -3 months
  For group T2x only.
Polynuclear basophils (g/l) | -4 months
  For group T2x only.
Polynuclear basophils (g/l) | -5 months
  For group T2x only.
Polynuclear basophils (g/l) | -6 months
  For group T2x only.
D-dimers (ng/ml) | -1 months
  For group T2x only.
D-dimers (ng/ml) | -2 months
  For group T2x only.
D-dimers (ng/ml) | -3 months
  For group T2x only.
D-dimers (ng/ml) | -4 months
  For group T2x only.
D-dimers (ng/ml) | -5 months
  For group T2x only.
D-dimers (ng/ml) | -6 months
  For group T2x only.
Fibrin monomers (ng/ml) | -1 months
  For group T2x only.
Fibrin monomers (ng/ml) | -2 months
  For group T2x only.
Fibrin monomers (ng/ml) | -3 months
  For group T2x only.
Fibrin monomers (ng/ml) | -4 months
  For group T2x only.
Fibrin monomers (ng/ml) | -5 months
  For group T2x only.
Fibrin monomers (ng/ml) | -6 months
  For group T2x only.
Trophoblast microparticles (%) | -1 months
  For group T2x only.
Trophoblast microparticles (%) | -2 months
  For group T2x only.
Trophoblast microparticles (%) | -3 months
  For group T2x only.
Trophoblast microparticles (%) | -4 months
  For group T2x only.
Trophoblast microparticles (%) | -5 months
  For group T2x only.
Trophoblast microparticles (%) | -6 months
  For group T2x only.
Angiogenic marker CD146 (ng/ml) | -1 months
  For group T2x only.
Angiogenic marker CD146 (ng/ml) | -2 months
  For group T2x only.
Angiogenic marker CD146 (ng/ml) | -3 months
  For group T2x only.
Angiogenic marker CD146 (ng/ml) | -4 months
  For group T2x only.
Angiogenic marker CD146 (ng/ml) | -5 months
  For group T2x only.
Angiogenic marker CD146 (ng/ml) | -6 months
  For group T2x only.
Total plasma concentration of nucleosomes (AU) | -1 months
  For group T2x only.
Total plasma concentration of nucleosomes (AU) | -2 months
  For group T2x only.
Total plasma concentration of nucleosomes (AU) | -3 months
  For group T2x only.
Total plasma concentration of nucleosomes (AU) | -4 months
  For group T2x only.
Total plasma concentration of nucleosomes (AU) | -5 months
  For group T2x only.
Total plasma concentration of nucleosomes (AU) | -6 months
  For group T2x only.
Total plasma concentration of free DNA (ng/ml) | -1 months
  For group T2x only.
Total plasma concentration of free DNA (ng/ml) | -2 months
  For group T2x only.
Total plasma concentration of free DNA (ng/ml) | -3 months
  For group T2x only.
Total plasma concentration of free DNA (ng/ml) | -4 months
  For group T2x only.
Total plasma concentration of free DNA (ng/ml) | -5 months
  For group T2x only.
Total plasma concentration of free DNA (ng/ml) | -6 months
  For group T2x only.
Fibrinogen (g/l) | Base line (day 0)
  For group P, baseline occurs within the 30 days preceding birth. For group T1, baseline = time of inclusion. For group T2, baseline occurs within the 30 days preceding birth.
Fibrinogen (g/l) | -1 months
  For group T2x only.
Fibrinogen (g/l) | -2 months
  For group T2x only.
Fibrinogen (g/l) | -3 months
  For group T2x only.
Fibrinogen (g/l) | -4 months
  For group T2x only.
Fibrinogen (g/l) | -5 months
  For group T2x only.
Fibrinogen (g/l) | -6 months
  For group T2x only.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Bouvier, MD, Study Director — Centre Hospitalier Universitaire de Nîmes; Eve Mousty, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Bouvier S, Mousty E, Fortier M, Demattei C, Mercier E, Nouvellon E, Chea M, Grosjean F, Letouzey V, Gris JC. Placenta-mediated complications: Nucleosomes and free DNA concentrations differ depending on subtypes. J Thromb Haemost. 2020 Dec;18(12):3371-3380. doi: 10.1111/jth.15105. Epub 2020 Oct 18. PMID 32979032
- [Derived] Bouvier S, Traboulsi W, Blois SM, Demattei C, Joshkon A, Mousty E, Nollet M, Paulmyer-Lacroix O, Foucault-Bertaud A, Fortier M, Leroyer AS, Bachelier R, Letouzey V, Alfaidy N, Dignat-George F, Blot-Chabaud M, Gris JC, Bardin N. Soluble CD146 is increased in preeclampsia and interacts with galectin-1 to regulate trophoblast migration through VEGFR2 receptor. F S Sci. 2022 Feb;3(1):84-94. doi: 10.1016/j.xfss.2021.11.002. Epub 2021 Nov 19. PMID 35559998